CLINICAL TRIAL: NCT05072938
Title: A Multi-center, Open-label, Randomized, Phase IV Clinical Trial to Compare the Efficacy and Safety of Rebamipide/Nizatidine Combination Therapy With Nizatidine Monotherapy in Patients With Gastritis
Brief Title: Clinical Trial to Compare Rebamipide/Nizatidine Combination Therapy With Nizatidine Monotherapy in Patients With Gastritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUC0S-P401
Record Dates: First submitted 2021-08-13; First posted 2021-10-11 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Gastritis
MeSH Terms: conditions — Gastritis | interventions — Nizatidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nizatidine Monotherapy (Active Comparator): Nizatidine Monotherapy
  Interventions: Drug: Axid Capsule 150mg
- Rebamipide/Nizatidine Combination Therapy (Experimental): Rebamipide/Nizatidine Combination Therapy
  Interventions: Drug: Mucotra SR Tablet 150mg

INTERVENTIONS:
Drug: Mucotra SR Tablet 150mg — Rebamipide/Nizatidine Combination Therapy
  Other Names: Mucotra
  Arms: Rebamipide/Nizatidine Combination Therapy
Drug: Axid Capsule 150mg — Nizatidine Monotherapy
  Other Names: Axid
  Arms: Nizatidine Monotherapy

SUMMARY:
The purpose of this study is to compare the Efficacy and Safety of Rebamipide/Nizatidine Combination Therapy with Nizatidine Monotherapy in Patients with Gastritis

DETAILED DESCRIPTION:
The purpose of this study is to compare the Efficacy and Safety of Rebamipide/Nizatidine Combination Therapy with Nizatidine Monotherapy in Patients with Gastritis.

Anticipated result is to prove superiority of Rebamipide/Nizatidine combination therapy at 2 weeks compared to Nizatidine Monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 19 years or older and under 75 years
2. Subject who was diagnosed with acute or chronic gastritis in upper gastrointestinal endoscopy conducted within 7 days prior to the start of administration of medications for clinical trials and identified at least one labyrinth (defect of mucosal surface layer)
3. Subject who voluntarily decides to participate in the trial after hearing the explanation of this clinical trial and signs the informed consent form.

Exclusion Criteria

1. Subject who is unable to examine the upper gastrointestinal endoscope
2. A person with the following past history

   * Surgery to suppress gastric acid secretion or gastrointestinal and esophagus surgery
   * Malignant tumor of the digestive system
   * overreacted to the components of medicine for clinical trials and H2 receptor blockers
   * Drug or alcohol abuse
3. A person accompanied by the following diseases

   * Digestive ulcers (excluding half a scar)
   * Reflux esophagitis
   * Inflammatory bowel disease (cron disease, ulcerative colitis)
   * Thrombotic diseases (such as cerebral thrombosis, myocardial infarction, thrombotic venous inflammation, etc.)
   * Zollinger-Ellison syndrome
   * Subject with mental illness, cardiovascular system, respiratory system, endocrine system, central nervous system who the investigator determined that it is difficult to participate in this clinical trial
4. A person who needs to administer a taboo drug during the clinical trial period.
5. Pregnant women and nursing women
6. Fertilized women and men who have a pregnancy plan or do not have the will to use the appropriate contraceptive method during the clinical trial period.
7. Subject with genetic problems such as galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption, etc.
8. Severe liver disorder (AST or ALT > 3 times the normal upper limit of the organ)
9. Serious nephropathy (creatinine clearance < 50 mL/min)
10. Subject who has been administered (applied) other clinical medications or medical devices within 4 weeks of screening
11. Subject who the investigator determined it is inappropriate to participate in this clinical trial.

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Effective rate of gastric mucosal erosion on the upper gastrointestinal endoscopy | 2 weeks
  Effective rate of gastric mucosal erosion on the upper gastrointestinal endoscopy at 2 weeks compated to baseline

SECONDARY OUTCOMES:
Erosion cure rate on upper gastrointestinal endoscopy | 2 weeks
  Erosion cure rate on upper gastrointestinal endoscopy at 2 weeks compared to baseline
Effective rate of bleeding on upper gastrointestinal endoscopy | 2 weeks
  Effective rate of bleeding on upper gastrointestinal endoscopy at 2 weeks compared to baseline
Effective rate of flares on upper gastrointestinal endoscopy | 2 weeks
  Effective rate of flares on upper gastrointestinal endoscopy at 2 weeks compared to baseline
Edema cure rate on upper gastrointestinal endoscopy | 2 weeks
  Edema cure rate on upper gastrointestinal endoscopy at 2 weeks compared to baseline
Validity rate of subjective symptom scores evaluated by subjects | 2 weeks
  Validity rate of subjective symptom scores evaluated by subjects at 2 weeks compared to baseline
Change in total subjective symptom score and individual symptom score assessed by the subject at 2 weeks compared to baseline | 2 weeks
  Change in total subjective symptom score and individual symptom score assessed by the subject

CONTACTS AND LOCATIONS:
Overall Officials: Myung Kyu Choi, Principal Investigator — The Catholic University of Korea
Locations (1):
- The Catholic University of Korea c St. Mary's Hospital, Seoul, South Korea